CLINICAL TRIAL: NCT00478738
Title: A Study to Assess the Pharmacokinetics of Single Escalating Doses of Inhaled GSK961081 DPI (a Dual Pharmacophore) in Healthy Subjects (Part 1) and a Randomised, Double-blind, Double Dummy, Crossover (Incomplete Block) Study to Assess the Safety, Tolerability, Pharmacodynamics (Pulmonary and Systemic) and Pharmacokinetics of 14 Days Dosing With Inhaled GSK961081 DPI Compared With Placebo and Tiotropium Plus Salmeterol in Patients With COPD (Part 2)
Brief Title: A 2 Part Study Examining Doses Of GSK961081 In Healthy Volunteers And Then In COPD Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MAB104958
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: b-agonist,; COPD.; pharmacodynamic,; pharmacokinetic,; anti muscarinic,
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — batefenterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK961081 (Other): GSK961081
  Interventions: Drug: GSK961081

INTERVENTIONS:
Drug: GSK961081

SUMMARY:
GSK961081 has previously been administered to healthy subjects in a nebulised formulation and the first part of this study which will be conducted in healthy subjects proposes to bridge the change from nebulised to DPI formulation of GSK961081 before administration to patients. The second part of the study will be conducted in COPD patients and aims to assess the safety and bronchodilator profile of GSK961081 over 24 hours, during 14 days dosing.

DETAILED DESCRIPTION:
A study to assess the pharmacokinetics of single escalating doses of inhaled GSK961081 DPI (a dual pharmacophore) in healthy subjects (Part 1) and a randomised, double-blind, double dummy, crossover (incomplete block) study to assess the safety, tolerability, pharmacodynamics (pulmonary and systemic) and pharmacokinetics of 14 days dosing with inhaled GSK961081 DPI compared with placebo and tiotropium plus salmeterol in patients with COPD (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female (of non-child bearing potential) > 40 years of age and < 75 years of age.
* Non- child bearing potential is defined as physiologically incapable of becoming pregnant, including females who are post menopausal ( more than 2 years without menses with appropriate clinical history ie age, history of vasomotor symptoms-estradiol and FSH levels may be checked if indicated) and females who are surgically sterile (hysterectomy, tubal ligation or bilateral oophorectomy.
* Subject diagnosed with COPD (stage II) in accordance with ATS/ERS guidelines (see Appendix 2: COPD Guidelines).
* Subject is a smoker or an ex smoker with a history of at least 10 pack years (1 pack year= 20 cigarettes smoked per day for 1 year or equivalent)
* Subject has FEV1/FVC < 0.7 post - bronchodilator (salbutamol)
* Subject has FEV1 < 80 % of predicted normal for height, age, gender after inhalation of salbutamol
* Response to ipratropium bromide defined as:

Either an increase in FEV1 of > 12 % and > 150 mLwithin 2 hour following inhalation of 80 µcg ipratropium bromide at the screening visit Or: a documented increase in FEV1 of >12 % and > 150 mL within 2 hour following inhalation of 80 µcg ipratropium bromide within 6 months of screening and an increase in FEV1 of > 6 % and > 100 mL within 2 h following inhalation of 80 mg ipratropium bromide at the screening visit (in order to allow for potential fluctuations in the response to ipratropium bromide in patients known to be responders to ipratropium bromide)

* Response to salbutamol defined as:

Either an increase in FEV1 of > 12 % and > 150 mL within 2 hour following inhalation of 400 mg salbutamol at the screening visit Or: a documented increase in FEV1 of >12 % and > 150 mL within 2 hour following inhalation of 400 mg salbutamol within 6 months of screening and an increase in FEV1 of > 6 % and >100 mL within 2 h following inhalation of 400 mg salbutamol at the screening visit (in order to allow for potential fluctuations in the response to salbutamol in patients known to be responders to salbutamol)

* Body mass index within the range 18-35 kilograms/metre² (kg/m²).
* Subject is able and willing to give written informed consent to take part in the study.
* Subject is available to complete all study measurements

Exclusion Criteria:

* Subjects who have a past or present disease, which as judged by the Investigator and medical monitor may affect the outcome of the study or the safety of the subject
* Women who are pregnant or lactating
* An unwillingness of subjects to abstain from sexual intercourse with pregnant or lactating women; or an unwillingness of the subject to use a condom/spermicide in addition to having their female partner use another form of contraception such as IUD, diaphragm with spermicide, oral contraceptives, injectable progesterone, subdermal implants or tubal ligation if the woman could become pregnant from the time of the first dose study medication until 90 days post-dose
* The subject has a positive urine drug screen. A minimum list of drugs that will be screened for include Amphetamines, barbiturates, Cocaine, Opiates, Cannabinoids and Benzodiazepines.
* The subject has a positive alcohol test (breath or urine) predose.
* A history, or suspected history, of alcohol abuse within the 6 months before the screening visit.
* A positive test for hepatitis C antibody, hepatitis B surface antigen, or HIV.
* The subject has participated in a clinical study with another New Chemical Entity within the past 2 months or a participated in a clinical study with any other drug during the previous month.
* The subject has donated a unit of blood within the 56 days or intends to donate within 56 days after completing the study.
* The subject has claustrophobia that may be aggravated by entering the plethysmography cabinet.
* Subject has an FEV1 < 50 % of predicted for age, height and gender after inhalation of salbutamol.
* The subject has a diagnosis of active tuberculosis, lung cancer, sarcoidosis, bronchiectasis, lung fibrosis, pulmonary hypertension or with a primary diagnosis of asthma
* The subject has a known allergy or hypersensitivity to ipratropium, salbutamol, tiotropium, salmeterol or lactose
* A subject in whom ipratropium, salbutamol, tiotropium and/or salmeterol is contraindicated
* Subjects with lung volume reduction surgery within 12 months of screening
* Poorly controlled COPD defined as:

Either: acute worsening of COPD that is managed by the subject at home by treatment with increased corticosteroids or antibiotics in the 6 weeks before screening Or: more than 2 exacerbations in the previous 12 months before screening that required a course of oral steroids or antibiotics, and/or required hospitalisation

* Subject has had a respiratory tract infection in the 4 weeks before screening
* Subject requires treatment with inhaled cromolyn sodium, theophyline, oral beta agonists, nebulised anticholinergics or leukotriene antagonists
* Subject is unable to abstain from long acting beta agonist from 72 hours before screening and throughout the dosing period
* Subject is unable to abstain from tiotropium from 28 days before screening and throughout the dosing period
* Subject is predicted to be unable to abstain from short acting inhaled beta agonists (to be used as rescue medication during the study) for 6 hours before screening and before study visits, when required, until all post dose lung function tests have been completed for a given study day.
* Subject has received oral corticosteroids within the 6 weeks before screening
* Subject is receiving > 1000 mg FP (or equivalent) a day of inhaled corticosteroid or has changed dose within the 6 weeks before screening or is predicted not to be able to maintain a constant dose during the study
* Subject is receiving oxygen therapy or nocturnal positive pressure treatment
* Subject has prostate hypertrophy or narrow angle glaucoma
* The subject is unable to use the dosing devices correctly.
* Subject with carcinoma that has not been in complete remission for at least 5 years (with the exception of carcinoma in situ of the cervix, squamous cell carcinoma and basal cell carcinoma if the subject is considered cured)
* A history of congestive heart failure, coronary insufficiency or cardiac arrhythmia
* Abnormal 12- lead ECG abnormality which is either clinically significant or may interfere with QTc measurement
* A supine mean heart rate outside the range 40-90 beats per minute (bpm) at screening.
* Elevated supine blood pressure higher than 160/95 at screening.
* Subject is receiving a diuretic and/ or beta adrenergic antagonist.
* Subject has a serum potassium level below the reference range at screening.
* Strict vegetarians;
* Shift-worker unable to comply with the study;
* Inability to understand the protocol requirements, instructions and study-related restrictions; the nature, scope and possible consequences of the study;
* Unlikely to complete the study; e.g., uncooperative attitude, inability to return for Follow-up Visits;
* Subject is the Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff, or relative thereof directly involved in the conduct of the study;
* Vulnerable individuals (e.g., persons kept in detention).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2007-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Part 1: Summary of area under the GSK961081 concentration-time curve (AUC) after a single dose | Pre-dose (0.0 hour [h]) and 15, 30, 45 minutes (M), 1, 2, 3, 4, 6, 8, 12 and 24 h post dose of each treatment period
  Plasma samples for PK analysis were drawn on Day (D) 1 at indicated time points. The AUC from time zero (0M) to 2h (AUC 0-2) was area under the plasma concentration-time curve over the 2h time period. AUC(0-6) was area under the plasma concentration-time curve from 0M to 6h. AUC(0-t) was area under the plasma concentration-time curve from 0M to last quantifiable concentration. The AUC extrapolated to infinity (inf) (AUC[0-inf]) was calculated as the sum of AUC(0-t) and Ct/lambda z, where Ct is the observed GSK961081 concentration obtained from the log-linear regression analysis of the last quantifiable time-point and lambda z is the terminal phase rate constant estimated by linear regression analysis of the log transformed concentration-time data. The number of time points used in the estimation of lambda z. Different participants may have been analyzed at different time points; thus, the overall number of participants analyzed reflects everyone in the PK population.
Part 1: Summary of maximum observed concentration (Cmax) of GSK961081 after a single dose | Pre-dose (0.0h) and 15, 30, 45 M, 1, 2, 3, 4, 6, 8, 12 and 24 h post dose of each treatment period
  Plasma samples for PK analysis were drawn on D1 at indicated time points. The first occurrence of the maximum observed GSK961081 concentration determined directly from the raw concentration-time data after each single dose. All participants were present at the time of measurement.
Part 1: Summary of last observed plasma concentration (t-last), time of maximum observed concentration (t-max) and terminal elimination half-life (t-half) | Pre-dose (0.0h) and 15, 30, 45 M, 1, 2, 3, 4, 6, 8, 12 and 24 h post dose of each treatment period
  Plasma samples for PK analysis were drawn on D1 at indicated time points. The t-last and t-max was determined directly from the raw concentration-time data after each single dose. The t-half was obtained as the ratio of ln2/lambda z, where ln(2) is the natural logarithm of 2 (approximately 0.693) and lambda z is the terminal phase rate constant estimated by linear regression analysis of the log transformed concentration-time data after each single dose. Data for adjusted mean is presented as least square mean. Only those participants available at the specified time points were analyzed (represented by n=x,x,x in the category titles). Different participants may have been analyzed at different time points; thus, the overall number of participants analyzed reflects everyone in the All Subjects population.
Part 2: Forced Expiratory Volume in 1 second (FEV1) over 24 hours post-dose on D1 and 14 | Up to D14 of each treatment period (up to 16 weeks)
  Lung function tests (FEV1) was recorded whilst the participant was in a sitting position (if taken whilst the participant was on the bed, their legs should be over the edge). All lung function tests was repeated, until three technically acceptable measurements were made. Each measurement should be done at least 1 M apart. Participants must be resting in the body box for at least 30 seconds prior to any assessments. The FEV1 was measured at 15, 30 M, 1, 4, 12 and 24 h post dose of each treatment period on D1 and 14. Data for adjusted mean is presented as least square mean. Only those participants available at the specified time points were analyzed (represented by n=x,x,x,x in the category titles). Different participants may have been analyzed at different time points; thus, the overall number of participants analyzed reflects everyone in the All Subjects population. Data for adjusted mean is presented as least square mean.

SECONDARY OUTCOMES:
Part 1: Number of participants with Adverse Events (AE) and Serious adverse events (SAE) | Up to 16 weeks
  An AE was defined as any untoward medical occurrence (MO) in a participant temporally associated with the use of a medicinal product (MP), whether or not considered related to the MP and can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with its use. The SAE was any untoward MO that, at any dose, results in death, life threatening, persistent or significant disability/incapacity, results in or prolongs inpatient hospitalization, congenital abnormality or birth defect, that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition. Refer to the general AE/SAE module for a list of AEs and SAEs.
Part 1: Mean values for urea, sodium, potassium, cholesterol, chloride, high density lipids-cholesterol (HDLC), and triglyceride | Up to D1 of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of indicated laboratory biochemistry tests on D1 pre-dose and 24h post dose in Part 1 of study. All participants were present at the time of measurement.
Part 1: Mean values for creatinine and total bilirubin | Up to D1of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of indicated laboratory biochemistry tests on D1 pre-dose and 24h post dose in Part 1 of study. All participants were present at the time of measurement.
Part 1: Mean values for total protein and albumin | Up to D1of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of indicated laboratory biochemistry tests on D1 pre-dose and 24h post dose in Part 1 of study. All participants were present at the time of measurement.
Part 1: Mean values for aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), creatine kinase and gamma glutamyl transferase (GGT). All participants were present at the time of measurement. | Up to D1of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of indicated laboratory biochemistry tests on D1 pre-dose and 24h post dose in Part 1 of study. All participants were present at the time of measurement.
Part 1: Mean values for platelet and white blood cell (WBC) | Up to D1 of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of indicated hematology tests on D1 pre-dose and 24h post dose in Part 1 of study.
Part 1: Mean values for hemoglobin and mean corpuscle hemoglobin concentration (MCHC) | Up to D1 of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of indicated hematology tests on D1 pre-dose and 24h post dose in Part 1 of study.
Part 1: Mean values for hematocrit | Up to D1 of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of indicated hematology tests on D1 pre-dose and 24h post dose in Part 1 of study.
Part 1: Mean values for mean corpuscle volume (MCV) | Up to D1 of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of indicated hematology tests on D1 pre-dose and 24h post dose in Part 1 of study.
Part 1: Mean values for mean corpuscle hemoglobin (MCH) | Up to D1 of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of indicated hematology tests on D1 pre-dose and 24h post dose in Part 1 of study.
Part 1: Mean values for reticulocytes, total neutrophil, lymphocyte, monocyte, eosinophil and basophil | Up to D1 of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of indicated hematology tests on D1 pre-dose and 24h post dose in Part 1 of study.
Part 1: Mean values for red blood cells (RBC) | Up to D1 of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of indicated hematology tests on D1 pre-dose and 24h post dose in Part 1 of study.
Part 1: Summary of Results of Statistical Serial Time point Analysis of FEV1 Data-Treatment Differences | Up to D1 of each treatment period (up to 16 weeks)
  Lung function tests (FEV1) was recorded whilst the participant was in a sitting position (if taken whilst the participant was on the bed, their legs should be over the edge). All lung function tests was repeated, until three technically acceptable measurements were made. Each measurement should be done at least 1 M apart. Participants must be resting in the body box for at least 30 seconds prior to any assessments. FEV1 measurements were taken after sGaw measurements. The FEV1 was measured at 15, 1, 4, 12 and 24 h post dose of each treatment period on D1. Data for adjusted mean is presented as least square mean. All participants were present at the time of measurement.
Part 1: Change from Baseline derived Electrocardiogram (ECG) parameters- QT interval corrected according to Bazzet's formula (QTcF) and QT interval corrected according to Fridericia's formula (QTcB) Maximum value (0-4 h) | Up to D1of each treatment period (up to 16 weeks)
  ECG measurements were made with the participants in a supine position having rested in this position for at least 10 M before each reading. Data is presented as maximum value 0-4 h of each treatment period on D1. The QTcB was derived automatically by the machine. The QTcF was manually derived by dividing QT interval with cube root of division of RR interval by 1000. Where, RR interval (milliseconds [msec]) was calculated as square of QT interval divided by QTcB, which was multiplied by 1000. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Baseline value was defined as the mean of the three pre-dose measurements on D1 for each treatment period. Data for adjusted mean is presented as least square mean.
Part 1: Change from Baseline derived ECG parameters-QTc(F) and QTc(B) Weighted mean (0-4 h)-Part | Up to D1 of each treatment period (up to 16 weeks)
  ECG measurements was made with the participants in a supine position having rested in this position for at least 10 M before each reading. The QTcB was derived automatically by the machine. The QTcF was manually derived by dividing QT interval with cube root of division of RR interval by 1000. Where, RR interval (msec) was calculated as square of QT interval divided by QTcB, which was multiplied by 1000. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Baseline value was defined as the mean of the three pre-dose measurements on D1 for each treatment period. All available data at the actual relative times were included in the derivation of the weighted mean with pre-dose measurements representing the time point zero, and all subsequent time points (0- 4 h) calculated relative to dosing in that period. Data for adjusted mean is presented as least square mean.
Part 1: Mean supine systolic blood pressure (SBP) maximum value (0-4 h) | Up to D1of each treatment period (up to 16 weeks)
  Participants were required to rest in the supine position for at least 10 M before each reading. SBP was measured with an automatic measuring device. Data is presented as maximum value 0-4 h of each treatment period on D1.Three baseline was defined as the mean of the three pre-dose measurements on D1 for each treatment period. Data for adjusted mean is presented as least square mean.
Part 1: Mean supine diastolic blood pressure (DBP) minimum change (0-4 h) | Up to D1 of each treatment period (up to 16 weeks)
  Participants were required to rest in the supine position for at least 10 M before each reading. DBP was measured with an automatic measuring device. Data is presented as minimum change 0-4 h of each treatment period on D1. The Baseline was defined as the mean of the three pre-dose measurements on D1 for each treatment period. Data for adjusted mean is presented as least square mean. Data for adjusted mean is presented as least square mean.
Part 1: Mean supine SBP and supine DBP Weighted mean (0-4 h) | Up to D1 of each treatment period (up to 16 weeks)
  Participants were required to rest in the supine position for at least 10 M before each reading. SBP and DBP were measured with an automatic measuring device. It was measured at 0- 4 h post dose of each treatment period on D1. The baseline was defined as the mean of the three pre-dose measurements on D1 for each treatment period. All available data at the actual relative times were included in the derivation of the weighted mean with pre-dose measurements representing the time point zero, and all subsequent time points calculated relative to dosing in that period. Data for adjusted mean is presented as least square mean.
Part 1: Change from Baseline supine heart rate maximum value (0-4 h) | Up to D1 of each treatment period (up to 16 weeks)
  Participants were required to rest in the supine position for at least 10 M before each reading. Heart rate was measured with an automatic measuring device. Data is presented as maximum value 0-4 h of each treatment period on D1. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. The baseline was defined as the mean of the three pre-dose measurements on D1 for each treatment period. Data for adjusted mean is presented as least square mean.
Part 1: Change from Baseline supine heart rate Weighted mean (0-4 h) | Up to D1 of each treatment period (up to 16 weeks)
  Participants were required to rest in the supine position for at least 10 M before each reading. Heart rate was measured with an automatic measuring device. It was measured at 0-4 h post dose of each treatment period on D1. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. The Baseline was defined as the mean of the three pre-dose measurements on D1 for each treatment period. All available data at the actual relative times were included in the derivation of the weighted mean with pre-dose measurements representing the time point zero, and all subsequent time points calculated relative to dosing in that period. Data for adjusted mean is presented as least square mean.
Part 1: Maximum change in postural SBP and DBP (0-4h) | Up to D1 of each treatment period (up to 16 weeks)
  Participants were required to rest in the supine position for at least 10 M before each reading. SBP and DBP were measured with an automatic measuring device. Data is presented as maximum value 0-4 h of each treatment period on D1. The Baseline was defined as the mean of the three pre-dose measurements on D1 for each treatment period. Maximum change in postural SBP and DBP (0-4 h) was derived as post dose standing reading minus post dose supine reading. Data for adjusted mean is presented as least square mean.
Part 1: Maximum change from Baseline value (0-4h) for glucose | Up to D1 of each treatment period (up to 16 weeks)
  Data is presented as maximum value of glucose at 0-4 h of each treatment period on D1. Blood samples were collected for measurement of glucose at pre-dose (0.0), 30 M, 1, 2 and 4 h post dose of each treatment period on D1. The Baseline was defined as the mean of the three pre-dose measurements on D1 for each treatment period. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Data for adjusted mean is presented as least square mean.
Part 1: Minimum change from Baseline value (0-4h) for potassium | Up to D1 of each treatment period (up to 16 weeks)
  Data is presented as minimum change for potassium at 0-4 h of each treatment period on D1. Blood samples were collected for measurement of potassium at pre-dose (0.0), 30 M, 1, 2 and 4 h post dose of each treatment period on D1. The Baseline was defined as the mean of the three pre-dose measurements on D1 for each treatment period. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Data for adjusted mean is presented as least square mean.
Part 1: Maximum change from Baseline value (0-4h) for potassium | Up to D1 of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of glucose at pre-dose (0.0), 30 M, 1, 2 and 4 h post dose of each treatment period on D1. The data for maximum change from Baseline for potassium was not analyzed.
Part 1: Weighted mean change from baseline (0-4h) for glucose and potassium | Up to D1 of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of glucose and potassium at pre-dose (0.0), 30 M, 1, 2 and 4 h post dose of each treatment period on D1. The Baseline was defined as the mean of the three pre-dose measurements on D1 for each treatment period. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. All available data at the actual relative times were included in the derivation of the weighted mean with pre-dose measurements representing the time point zero, and all subsequent time points calculated relative to dosing in that period. Data for adjusted mean is presented as least square mean.
Part 1: Number of participants with abnormal Holter ECG findings as a function of cardiac monitoring | Up to D1 of each treatment period (up to 16 weeks)
  Holter monitoring (24 h) was conducted at screening and after each dose during. Holter tapes were analyzed locally at site. A screening visit was taken place within 28 days of the first dosing occasion. Participants with abnormal (not clinically significant [NCS]), abnormal (clinically significant [CS]) and no result were presented.
Part 1: Number of participants with abnormal Lead II ECG findings as a function of cardiac monitoring | Up to D1 of each treatment period (up to 16 weeks)
  Lead II ECG monitoring (via telemetry) will be recorded from pre-dose until 6 h after the dose. Participants with abnormal (NCS), abnormal (CS) and no result were presented.
Part 2: Number of participants with AE and SAE | Up to 16 weeks
  An AE was defined as any untoward MO in a participant temporally associated with the use of a MP, whether or not considered related to the MP and can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with its use. The SAE was any untoward MO that, at any dose, results in death, life threatening, persistent or significant disability/incapacity, results in or prolongs inpatient hospitalization, congenital abnormality or birth defect, that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition. Refer to the general AE/SAE module for a list of AEs and SAEs.
Part 2: Mean values for urea, sodium, potassium, cholesterol, chloride, high density lipids-cholesterol (HDLC), and triglyceride | Up to D14 of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of indicated laboratory biochemistry tests on D1, 4, 7, 14 pre-dose and 24h post dose on D14 in Part 2 of study.
Part 2: Mean values for creatinine and total bilirubin | Up to D14 of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of indicated laboratory biochemistry tests on D1, 4, 7, 14 pre-dose and 24h post dose on D14 in Part 2 of study.
Part 2: Mean values for total protein and albumin | Up to D14 of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of indicated laboratory biochemistry tests on D1, 4, 7, 14 pre-dose and 24h post dose on D14 in Part 2 of study.
Part 2: Mean values for AST, ALT, ALP, creatine kinase and GGT | Up to D14 of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of indicated laboratory biochemistry tests on D1, 4, 7, 14 pre-dose and 24h post dose on D14 in Part 2 of study.
Part 2: Mean values for hemoglobin and MCHC | Up to D14 of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of indicated laboratory biochemistry tests on D1, 4, 7, 14 pre-dose and 24h post dose on D14 in Part 2 of study.
Part 2: Mean values for hematocrit | Up to D14 of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of indicated laboratory biochemistry tests on D1, 4, 7, 14 pre-dose and 24h post dose on D14 in Part 2 of study.
Part 2: Mean values for MCV | Up to D14 of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of indicated laboratory biochemistry tests on D1, 4, 7, 14 pre-dose and 24h post dose on D14 in Part 2 of study.
Part 2: Mean values for MCH | Up to D14 of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of indicated laboratory biochemistry tests on D1, 4, 7, 14 pre-dose and 24h post dose on D14 in Part 2 of study.
Part 2: Mean values for total neutrophil, lymphocyte, monocyte, eosinophil and basophil | Up to D14 of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of indicated laboratory biochemistry tests on D1, 4, 7 pre-dose and 24h post dose on D14 in Part 2 of study.
Part 2: Mean values for platelets and WBC | Up to D14 of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of indicated laboratory biochemistry tests on D1, 4, 7, 14 pre-dose and 24h post dose on D14 in Part 2 of study.
Part 2: Mean values for RBC | Up to D14 of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of indicated laboratory biochemistry tests on D1, 4, 7, 14 pre-dose and 24h post dose on D14 in Part 2 of study.
Part 2: Mean values for reticulocytes | Up to D14 of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of indicated laboratory biochemistry tests on D1, 4, 7 pre-dose and 24h post dose on D14 in Part 2 of study.
Part 2: Change from Baseline derived ECG parameters- QTcF and QTcB Maximum value (0-4 h) | Up to D14 of each treatment period (up to 16 weeks)
  ECG measurements were made with the participants in a supine position having rested in this position for at least 10 M before each reading. Data is presented as maximum value of glucose at 0-4 h of each treatment period on D1 and D14. The QTcB was derived automatically by the machine. The QTcF was manually derived by dividing QT interval with cube root of division of RR interval by 1000. Where, RR interval (msec) was calculated as square of QT interval divided by QTcB, which was multiplied by 1000. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Baseline value was defined as the mean of the three pre-dose measurements on D1 for each treatment period. Data for adjusted mean is presented as least square mean.
Part 2: Change from Baseline derived ECG parameters-QTcF and QTcB Weighted mean (0-4 h) | Up to D14 of each treatment period (up to 16 weeks)
  ECG measurements was made with the participants in a supine position having rested for at least 10 M before reading. Data is presented as maximum value of glucose at 0-4 h of each treatment period on D1 and D14. The QTcB was derived automatically by the machine. The QTcF was manually derived by dividing QT interval with cube root of division of RR interval by 1000. Where RR interval (msec) was calculated as square of QT interval divided by QTcB, which was multiplied by 1000. The change from Baseline was calculated by subtracting the Baseline values from the post-randomization values. Baseline value was defined as the mean of three pre-dose measurements on D1 for each treatment period. All available data at the actual relative times were included in the derivation of the weighted mean with pre-dose measurements representing the time point zero, and all subsequent time points (0-4 h) calculated relative to dosing in that period. Data for adjusted mean is presented as least square mean.
Part 2: Maximum change from Baseline value (0-4h) for potassium | Up to D14 of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of glucose at pre-dose (0.0), 30 M, 1, 2 and 4 h post dose of each treatment period on D1 and D14. The data for maximum change from Baseline was not analyzed.
Part 2: Ambulatory blood pressure: maximum, minimum, time to maximum, time to minimum and weighted mean for systolic and diastolic blood pressure, and weighted mean arterial pressure over 0-8 and 8-24 h after dosing on Days 1 and 14 | Up to D14 of each treatment period (up to 16 weeks)
  Ambulatory blood pressure was monitored over 0-8 h and 8-24 h after dosing of each treatment period on D1 and D14. The data for ambulatory blood pressure was not analyzed.
Part 2: Number of participants with abnormal Holter ECG findings as a function of cardiac monitoring | Up to D14 of each treatment period (up to 16 weeks)
  Holter monitoring (24 h) was conducted at screening and on D1 and 14 of each treatment period. Holter tapes were analyzed locally at site. A screening visit was taken place within 28 days of the first dosing occasion. Participants with abnormal (not clinically significant), abnormal (clinically significant) and no result were presented.
Part 2: Number of participants with abnormal Lead II ECG findings as a function of cardiac monitoring | Up to D14 of each treatment period (up to 16 weeks)
  Lead II ECG monitoring (via telemetry) will be recorded from pre-dose until 8 h after the dose on D1 and D14 of each treatment period. Participants with abnormal (not clinically significant), abnormal (CS) and no result were presented.
Part 2: Mean supine SBP maximum value (0-4 h) | Up to D14 of each treatment period (up to 16 weeks)
  Participants were required to rest in the supine position for at least 10 M before each reading. SBP was measured with an automatic measuring device. Data is presented as maximum value 0-4 h of each treatment period on D1 and D14. The baseline was defined as the mean of the three pre-dose measurements on D1 and D14 for each treatment period. Data for adjusted mean is presented as least square mean.
Part 2: Mean supine DBP minimum change (0-4 h) | Up to D14 of each treatment period (up to 16 weeks)
  Participants were required to rest in the supine position for at least 10 M before each reading. DBP was measured with an automatic measuring device. Data is presented as minimum change 0-4 h of each treatment period on D1 and D14. The baseline was defined as the mean of the three pre-dose measurements on D1 for each treatment period. Data for adjusted mean is presented as least square mean. Data for adjusted mean is presented as least square mean.
Part 2: Mean supine SBP and supine DBP Weighted mean (0-4 h) | Up to D14 of each treatment period (up to 16 weeks)
  Participants were required to rest in the supine position for at least 10 M before each reading. SBP and DBP were measured with an automatic measuring device. It was measured at 0- 4 h post dose of each treatment period on D1 and D14. The baseline was defined as the mean of the three pre-dose measurements on D1 for each treatment period. All available data at the actual relative times were included in the derivation of the weighted mean with pre-dose measurements representing the time point zero, and all subsequent time points calculated relative to dosing in that period. Data for adjusted mean is presented as least square mean.
Part 2: Change from Baseline supine heart rate maximum value (0-4 h) | Up to D14 of each treatment period (up to 16 weeks)
  Participants were required to rest in the supine position for at least 10 M before each reading. Heart rate was measured with an automatic measuring device. Data is presented as maximum value 0-4 h of each treatment period on D1 and D14. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. The baseline was defined as the mean of the three pre-dose measurements on D1 for each treatment period. Data for adjusted mean is presented as least square mean.
Part 2: Change from Baseline supine heart rate Weighted mean (0-4 h) | Up to D14 of each treatment period (up to 16 weeks)
  Participants were required to rest in the supine position for at least 10 M before each reading. Heart rate was measured with an automatic measuring device. It was measured at 0-4 h post dose of each treatment period on D1 and D14. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. The Baseline was defined as the mean of the three pre-dose measurements on D1 for each treatment period. All available data at the actual relative times were included in the derivation of the weighted mean with pre-dose measurements representing the time point zero, and all subsequent time points calculated relative to dosing in that period. Data for adjusted mean is presented as least square mean.
Part 2: Maximum change in postural SBP and DBP (0-4h) | Up to D14 of each treatment period (up to 16 weeks)
  Participants were required to rest in the supine position for at least 10 M before each reading. SBP and DBP were measured with an automatic measuring device. Data is presented as maximum value 0-4 h of each treatment period on D1 and D14. The Baseline was defined as the mean of the three pre-dose measurements on D1 for each treatment period. Maximum change in postural SBP and DBP (0-4h) was derived as post dose standing reading minus post dose supine reading. Data for adjusted mean is presented as least square mean.
Part 2: Minimum change from Baseline value (0-4h) for potassium | Up to D14 of each treatment period (up to 16 weeks)
  Data is presented as minimum change for potassium at 0-4 h of each treatment period on D1 and D14. Blood samples were collected for measurement of potassium at pre-dose (0.0), 30 M, 1, 2 and 4 h post dose of each treatment period on D1 and D14. The Baseline was defined as the mean of the three pre-dose measurements on D1 for each treatment period. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. Data for adjusted mean is presented as least square mean.
Part 2: Weighted mean change from baseline (0-4h) for potassium | Up to D14 of each treatment period (up to 16 weeks)
  Blood samples were collected for measurement of glucose and potassium at pre-dose (0.0), 30 M, 1, 2 and 4 h post dose of each treatment period on D1 and D14. The Baseline was defined as the mean of the three pre-dose measurements on D1 for each treatment period. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. All available data at the actual relative times were included in the derivation of the weighted mean with pre-dose measurements representing the time point zero, and all subsequent time points calculated relative to dosing in that period. Data for adjusted mean is presented as least square mean.
Part 2: Summary of AUC after a single dose | Pre-dose (0.0 h) and 30 M, 1, 2, 4, 6, 8, 12 and 24 h post dose of each treatment period on D1 and D14; Pre-dose (0.0 h) and 30 M, 1, 2, 4 and 6 h post dose of each treatment period on D7.
  Plasma samples for PK analysis were drawn on D1, 7 and 14 at indicated time points of each treatment period. The AUC from time zero (0M) to 2h (AUC 0-2) was area under the plasma concentration-time curve over the 2h time period. AUC(0-6) was area under the plasma concentration-time curve from 0M to 6h. AUC(0-t) was area under the plasma concentration-time curve from 0M to last quantifiable concentration. The AUC extrapolated to inf (AUC[0-inf]) was calculated as the sum of AUC(0-t) and Ct/lambda z, where Ct is the observed GSK961081 concentration obtained from the log-linear regression analysis of the last quantifiable time-point and lambda z is the terminal phase rate constant estimated by linear regression analysis of the log transformed concentration-time data. The number of time points used in the estimation of lambda z.
Part 2: Summary of Cmax of GSK961081 after a single dose | Pre-dose (0.0 h) and 30 M, 1, 2, 4, 6, 8, 12 and 24 h post dose of each treatment period on D1 and D14; Pre-dose (0.0 h) and 30 M, 1, 2, 4 and 6 h post dose of each treatment period on D7.
  Plasma samples for PK analysis were drawn on D1, 7 and 14 at indicated time points of each treatment period. The first occurrence of the maximum observed GSK961081 concentration determined directly from the raw concentration-time data after each single dose. All participants were present at the time of measurement.
Part 2: Summary of t-last, t-max and t-half | Pre-dose (0.0 h) and 30 M, 1, 2, 4, 6, 8, 12 and 24 h post dose of each treatment period on D1 and D14; Pre-dose (0.0 h) and 30 M, 1, 2, 4 and 6 h post dose of each treatment period on D7.
  PK population. Only those participants available at the specified time points were analyzed (represented by n=x,x in the category titles). Different participants may have been analyzed at different time points; thus, the overall number of participants analyzed reflects everyone in the PK population.
Part 2: Serial sGaw measurement over 24 hours post-dose on D1 and 14 | Up to D14 of each treatment period (up to 16 weeks)
  sGaw was assessed by whole body plethysmography at 30 M, 1, 4, 12 and 24 h post dose of each treatment period on D1 and D14. Participants must be resting in the body box for at least 30 seconds prior to any assessments. Data for adjusted

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Germany (2):
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Berlin, State of Berlin
- South Africa (3):
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, George
  - GSK Investigational Site, Mowbray

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bateman ED, Kornmann O, Ambery C, Norris V. Pharmacodynamics of GSK961081, a bi-functional molecule, in patients with COPD. Pulm Pharmacol Ther. 2013 Oct;26(5):581-7. doi: 10.1016/j.pupt.2013.03.015. Epub 2013 Mar 26. PMID 23538170
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: MAB104958 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: MAB104958 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: MAB104958 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: MAB104958 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: MAB104958 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: MAB104958 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: MAB104958 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register